CLINICAL TRIAL: NCT05654220
Title: A Randomized Controlled Trial to Link Emergency Department Patients to Navigation Services for Enrollment in Public Benefits
Brief Title: Linking Emergency Department Patients to Assistance Programs Study
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Benefits Data Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 852553
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Social Determinants of Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control (No Intervention): Participants in the control group will receive a summary flyer providing contact information for benefits enrollment navigators at BenePhilly, which includes a unique study phone line provided by Benefits Data Trust. Currently, the standard of care is for ED patients to receive no information about public benefits. Therefore, the flyer represents an augmentation of usual care for patients randomized to the control group.
- Intervention (Experimental): Participants in the intervention arm will receive a summary flyer providing contact information for benefits enrollment navigators at BenePhilly and will be instructed that study personnel will contact them one-day post-discharge to help connect them to a BDT enrollment navigator to help them submit their applications for public benefits. At Day 1 post-discharge, participants in the intervention group will receive a text message to prompt them to call the BDT enrollment navigators to complete their applications for public benefits they screened for while in the ED. On Day 3, patients will receive a follow-up message to assess whether they have contacted BDT. Those participants who indicate they have not yet connected with BDT on Day 3 will receive reminder text messages at Day 7 and 14 post-discharge.
  Interventions: Behavioral: Text Messaging Intervention

INTERVENTIONS:
Behavioral: Text Messaging Intervention — A text messaging intervention will be conducted that includes prompts to call trained BenePhilly enrollment specialists to submit applications for benefits programs. Text message prompts will be sent on days 2, 4, 7, 14, and 21 post-discharge from a Penn Medicine emergency department.
  Arms: Intervention

SUMMARY:
The objective of this randomized controlled trial is to test the effect of screening patients in Penn Medicine Emergency Departments for eligibility of public benefits programs and using text messages post-discharge to connect patients to benefits enrollment specialists at Benefits Data Trust (BDT). Eligible patients will be randomly selected to receive text messages for two weeks after Emergency Department discharge with the phone number to speak with a benefits enrollment specialist at BDT. The number of calls to the BDT phone line and the number of submitted applications to public benefits programs will be compared between patients receiving a summary flyer with the phone number for BDT and the text message intervention to connect with BDT in comparison to an active control group who receives only a summary flyer with the phone number for BDT.

DETAILED DESCRIPTION:
Every year, Philadelphians fail to claim approximately $450 million dollars in federal and state benefits1. Across the United States, unclaimed benefits are estimated at approximately $60 billion1. These benefits include support for food, housing, healthcare, economic support, and others that can make a significant impact on well-being, upward mobility, and financial stability. The reasons that benefits are unclaimed are numerous, including lack of awareness about benefit programs and eligibility criteria, lack of agency and self-efficacy in completing expansive application requirements and organizing the necessary paperwork, and navigating the psychological costs of stigma associated with seeking public benefits2. In accordance with incentive structures developed as a result of the Affordable Care Act, health care systems have demonstrated value in screening for patients' social needs and creating partnerships with public service agencies to connect patients to social services to improve individual and population health and reduce health care disparities3-5. Patients presenting to emergency departments are more likely to possess unmet social needs6-8. Thus, it is critical for health care providers in emergency departments to effectively identify patients' social needs and connect patients to social services agencies that can provide both immediate and long-term assistance through the connection to public benefits programs.

Benefits Data Trust (BDT), a benefits support organization based in Philadelphia, has a long track record of success in consistently securing benefits for individuals with unmet social needs. BDT assists individuals with the completion and submission of applications for 19 public benefits programs (e.g., Supplemental Nutrition Assistance Program, the Low-Income Home Energy Assistance Program, and the Pharmaceutical Contract for the Elderly) via different channels, including web, phone, text, and in-person support services. Trained outreach specialists are knowledgeable about the intricacies of benefits applications and eligibility requirements, and support is available in multiple languages. Building trust with clients and serving vulnerable underserved communities is a central focus for outreach specialists. For services that they do not provide assistance for, BDT is also staffed to provide warm handoffs to help connect individuals to relevant organizations.

The focus of this proposal is to test whether patients identified in Penn Medicine Emergency Departments (ED) randomized to receive a warm handoff text messaging intervention are more likely to connect to study-specific BDT phone line and submit more applications for public benefits programs in comparison to patients who only receive a summary flyer with the BDT study-specific phone line upon discharge from the Emergency Department.

We will first conduct a pilot study with 30 participants to assess the design efficacy and implementation success of the text messaging intervention. After which, we will concurrently launch a two-arm prospective intervention randomized controlled trial that is expected to occur over 6 months in Penn Medicine Emergency Departments. The study will use Way To Health, a research information technology platform at the University of Pennsylvania used previously in digital health engagement clinical trials.

We propose to first survey patients to determine their eligibility for public benefits programs. Second, patients who are eligible for at least 1 of the 21 benefits programs to which BDT either provides direct application support or provides referrals to agency websites to complete applications will be randomly selected to either receive a flyer with the study-specific BDT phone number to apply for public benefits programs (active control) or receive a text messaging intervention for two weeks after leaving the ED with instructions to connect to the BDT study-specific phone line in addition to the flyer. Patients randomized to the intervention arm will receive an initial text message one-day post-discharge from the ED with instructions for connecting with BDT and will receive subsequent reminders to connect with BDT on Days 3, 7, and 14 post-discharge. Patients who indicate that they have successfully connected with BDT on Day 3 will not receive intervention messages on Days 7 and 14. All patients, both those randomized to the control and intervention groups, will receive an end-of-study survey on Day 14 post-discharge from the ED to ask patients if they connected with BDT, assess the patient's experience in the research study, and provide a reminder about the number to connect with BDT.

Insights from this randomized controlled trial will inform future work evaluating benefits enrollment outcomes, the relationship between benefits enrollment and health care outcomes, and variations in health services use among patients connected to BDT in the ED.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study based on the following criteria:

* Adults at least 18 years of age
* Patients must legally reside in Philadelphia
* Patients receiving care from Penn Medicine Emergency Departments at the Hospital of the University of Pennsylvania and Penn Presbyterian Medical Centerwho are deemed unlikely to require inpatient hospitalization or observation at the time of enrollment
* Patients must have one of the following insurance plans: Medicaid and/or Medicare (managed and traditional).
* Patient must be able to read/write in English.
* Patients must be eligible for at least 1 of the benefits programs for which BDT can provide either direct application assistance or provide a referral to the social services agency website to submit applications.
* Patients have a stable mobile phone number for the next 3 weeks.

Exclusion Criteria:

Patients will be excluded from participating in the study based on the following criteria:

* Individuals < 18 years
* Patients deemed by ED physicians to be in critical or unstable condition
* Does not speak/read English
* Patient is in severe distress, e.g., respiratory, physical, or emotional distress
* Patient is intoxicated, unconscious, or unable to appropriately respond to questions
* Patients under police custody
* Patients with a positive COVID-19 test
* Patients with private health insurance benefits or without health insurance
* Patients without a stable mobile phone number for the next 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Participant Connection to BDT | 14 days post-discharge from the emergency department
  Participant connection to BDT measured by phone calls completed by confirmed participants to BDT.

SECONDARY OUTCOMES:
Number of Applications Submitted | 14 days post-discharge from the emergency department
  Number of applications for public benefits programs submitted per participant by BDT.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Kilaru, MD, MSHP, Principal Investigator — Principal Investigator
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilaru AS, Haider A, Harrison J, Dixon EL, Southwick L, Berkowitz M, Rareshide C, Carroll C, Kaledin C, McDermott G, Mehta M, Stephens Shields AJ, De La Rosa W, Agarwal AK, Merchant RM. Linkage of Emergency Department Patients With Public Benefits Navigators via Text Messages: A Randomized Clinical Trial. JAMA Health Forum. 2026 Feb 6;7(2):e256637. doi: 10.1001/jamahealthforum.2025.6637. PMID 41649829